CLINICAL TRIAL: NCT04289909
Title: Identification of Retinal Perivascular Inflammation in Patients With Multiple Sclerosis Using Adaptive Optics
Brief Title: Identification of Retinal Perivascular Inflammation in Patients With Multiple Sclerosis Using Adaptive Optics (RETIMUS)
Acronym: RETIMUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C19-25
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Relapsing Remitting Multiple Sclerosis; Progressive Multiple Sclerosis; Optic Neuritis; Eye Diseases; Optic Nerve Diseases; Nervous System Diseases; Multiple Sclerosis
Keywords: relapsing remitting Multiple sclerosis; Progressive Multiple Sclerosis; Optic neuritis; multiple sclerosis; adaptive optics; eye disease; peripheral nervous system disease
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Optic Neuritis; Eye Diseases; Optic Nerve Diseases; Nervous System Diseases; Multiple Sclerosis; Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MS patients (Other): RRMS Patients with optic neuritis, RRMS patients without optic neuritis or Progressive MS patients
  Interventions: Other: Adaptive Optics Ophthalmoscopy (AOO)
- Control group (Other): Healthy volunteers
  Interventions: Other: Adaptive Optics Ophthalmoscopy (AOO)

INTERVENTIONS:
Other: Adaptive Optics Ophthalmoscopy (AOO) — AOO will permit to detect and quantify retinal perivascular inflammation in patients with MS in comparison to Healthy volunteers (control group)

SUMMARY:
Using a technique called adaptive optics imaging applied on retina, investigators aim to gain access to vascular changes that could occur early in the course of Multiple Sclerosis (MS) and which could reflect vascular changes occurring along the optic nerve of the brain parenchyma. Indeed, our team has been able to develop a quantitative method to measure the perivascular infiltrate in the retina of patients with various inflammatory retinal disease. It has been observed in MS patients that this perivascular infiltrate can also be detected in the retina. However, its distribution across MS phenotypes (relapsing or progressive MS, with and without optic neuritis) is still unknown.

DETAILED DESCRIPTION:
This is a monocentric pathophysiological, interventional, prospective, open label, non-randomized pilot study which aims to identify in patients with MS at different stages if the presence of retinal perivascular inflammation can be detected and quantified using adaptive optics, which is a non-invasive examination.

Investigators will recruit MS patients in 3 subgroups, depending on their phenotype (Relapsing Remitting Multiple Sclerosis (RRMS) without optic neuritis, RRMS with optic neuritis, progressive MS), with 15 patients in each group.

15 healthy volunteers (HV) will also be enrolled.

The comparison of these groups is necessary to determine if there are significant differences, allowing us to highlight biomarkers in MS patients in order to enable highly efficient and robust trials designs in the future.

To test the hypothesis, the study has 3 visits over 6 months (M0, M3 and M6). Neurological evaluation, blood sample, imaging, ophthalmologic evaluation and Adaptive optics ophthalmoscopy assessments will be performed.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* Age between 18 and 60 years old.
* Relapsing remitting MS (criteria of McDonald 2017)
* Less than 10 years of disease duration
* Subject who has never presented a clinical episode of optic neuritis
* Affiliation to a social security scheme or beneficiary of such a scheme

Group 2:

* Age between 18 and 60 years old
* Relapsing remitting MS (criteria of McDonald 2017)
* Less than 10 years of disease duration
* Subject presenting an acute episode of retrobulbar optic neuritis within 3 months from onset
* After optimal treatment for the retrobulbar optic neuritis
* Affiliation to a social security scheme or beneficiary of such a scheme

Group 3:

* Age between 18 and 60 years old
* Primary or Secondary progressive multiple sclerosis within 10 years of progressive phase;
* Affiliation to a social security scheme or beneficiary of such a scheme

Group 4 (Healthy Subjects):

* Age between 18 and 60 years old
* Affiliation to a social security scheme or beneficiary of such a scheme

Exclusion Criteria:

For all patients (Group 1; 2; 3):

* Corticosteroid treatment within one month from inclusion
* Other neurological, ophthalmologic or systemic disease;
* Severe symptoms of uncontrolled chronic disease (renal, hepatic, hematologic, gastro-intestinal, pulmonary or cardiac or any intercurrent uncontrolled disease at inclusion)
* Severe renal dysfunction (glomerular filtration rate < 30mL/min). This non-inclusion criteria will be verified by serum creatinine test within six months from inclusion;
* Contraindication for MRI;
* Pregnancy or breast-feeding;
* Unwillingness to be informed in case of abnormal MRI (with a significant medical anomaly)
* Incapacity to understand or sign the consent form;
* Adults legally protected (under judicial protection, guardianship, or supervision), persons deprived of their liberty.

For healthy subjects (Group 4):

* Neurological, ophthalmologic or systemic disease;
* Severe symptoms of uncontrolled chronic disease (renal, hepatic, hematologic, gastro-intestinal, pulmonary or cardiac or any intercurrent uncontrolled disease at inclusion);
* Contraindication for MRI;
* Pregnancy or breast-feeding;
* Unwillingness to be informed in case of abnormal MRI (with a significant medical anomaly)
* Incapacity to understand or sign the consent form;
* Adults legally protected (under judicial protection, guardianship, or supervision), persons deprived of their liberty.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Quantification of retinal perivascular cuff width across MS phenotypes | Baseline
  The primary endpoint is to quantify retinal perivascular cuff width across MS phenotypes, compared among a group of control at baseline.

SECONDARY OUTCOMES:
Variation of size of perivascular sheathing | month 3 and month 6
  Variation of size of perivascular sheathing along retinal vessels in the posterior pole during follow up (at month 3 and month 6) in patients with MS and a group of control
Clinical disability measure with EDSS | month 3 and month 6
  Evolution of Clinical disability: Expanded Disability Status Scale (EDSS: 0: normal neurological exam; 10 : death of the patient) at month 3 for MS patients with optic neuritis and at month 6 for all MS patients
Clinical disability measured with MSFC | month 3 and month 6
  Evolution of Clinical disability: Multiple Sclerosis Functional Composite (MSFC) at month 3 for MS patients with optic neuritis and at month 6 for all MS patients
Number of relapses | month 3 and month 6
  Evolution of Clinical disability: number of relapses at month 3 for MS patients with optic neuritis and at month 6 for all MS patients
Presence of disc oedema measured at Optical Coherence Tomography (OCT) measurements | month 3 and month 6
  Evolution of OCT measurements (presence of disc oedema) at month 3 for MS patients with optic neuritis and at month 6 for all MS patients
RNLF thickness measured at Optical Coherence Tomography (OCT) measurements | month 3 and month 6
  Evolution of OCT measurements : retinal nerve fiber layer thickness (RNFL, µm) at month 3 for MS patients with optic neuritis and at month 6 for all MS patients
parenchymal T2 lesion volume at MRI | Baseline
  Evolution of MRI metrics: parenchymal T2 lesion volume
gadolinium enhanced T1 lesion at MRI | Baseline
  Evolution of MRI metrics: gadolinium enhanced T1 lesion
optic nerve cross-sectional area at MRI | Baseline
  Evolution of MRI metrics: optic nerve cross-sectional area
Hyperintensity on the optic nerve at MRI | Baseline
  Evolution of MRI metrics: Hyperintensity on the optic nerve

CONTACTS AND LOCATIONS:
Overall Officials: Celine Louapre, MD, PHD, Principal Investigator — Institut du Cerveau et de la Moelle Epinière
Locations (1):
- Institut du Cerveau et de la Moelle epiniere - Hopital Pitie Salpetriere, Paris, France